CLINICAL TRIAL: NCT02468570
Title: A Phase 3 Substudy to Evaluate Executive Function in Adults With Phenylketonuria Who Are Participating in the Phase 3 Study, 165-302
Brief Title: A Phase 3 Substudy to Evaluate Executive Function in Adults With PKU Who Are Participating in the Phase 3 Study, 165-302
Acronym: PRISM303
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 165-303
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Phenylketonuria
Keywords: PKU; PEG-PAL; Pegvaliase; BMN 165; rAv-PAL PEG; PRISM 302; PRISM 303; BioMarin; 165-302
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Administration of CANTAB and Subject Global Assessment — At designated visits, subject will perform the CANTAB tasks and complete the Subject Global Assessment Questionnaire

SUMMARY:
A Phase 3 substudy to evaluate executive function in adults with phenylketonuria who are participating in the phase 3 Study, 165-302. Approximately 100 subjects, aged ≥ 18 to ≤ 70 years old, with PKU will be enrolled.

DETAILED DESCRIPTION:
Study 165-303, is a Phase 3 substudy enrolling approximately 100 subjects, aged ≥ 18 to ≤ 70 years old, with PKU who are participating in the Phase 3 study, 165-302.

Per the 165-303 protocol, the investigator does not assign a specific intervention to the study participants. In accordance with the protocol for Study 165-303, subjects were asked to perform selected set of three tasks from the CANTAB tool (Rapid Visual Processing [RVP], Spatial Working Memory [SWM], and Stop Signal Task [SST]) to assess executive function and each subject's self perception of their current state was measured using a subject global assessment questionnaire that contains seven questions about current state perception of attention, energy level, tiredness, confusion, sadness, anger and tension.

The time points for administering the above tools are as follows, which coincide with time points in part 2 and part 4 of Study 165-302: screening (entry into Part 2 165-302 Day 1 of Week 1), baseline visit (Part 2 Week 8), and 3 additional study visits at different time points in the Part 4 of 165-302 study.

ELIGIBILITY:
Inclusion Criteria:

* Are currently participating in Part 1 of Study 165-302 and meet the criteria for participation in Part 2 of 165-302
* Are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures.
* Have the ability to complete the CANTAB and subject global assessment.
* Are willing and able to comply with all study procedures.

Exclusion Criteria:

* Any condition that, in the view of the investigator, places the subject at high risk of poor compliance or terminating early from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with PKU who are currently enrolled in 165-302 Part 2.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lounsbury, Study Director — Principal Scientist/Medical Monitor
Locations (4):
- United States (4):
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BioMarin Pharmaceutical Website — http://www.bmrn.com
- See also: BioMarin sponsored PKU educational/community website — http://www.pku.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pooled Results: This is a sub-study of 165-302, with a randomized, placebo-control discontinuation design in Part 2. 9 subjects were enrolled in 165-303: 3 in 20mg/day and 3 in 40mg/day Active arm, 2 in 20mg/day and 1 in 40mg/day Placebo arm. Data interpretability was extremely limited, hence planned analysis was using the pooled treatment groups.
Groups:
- Pooled Active: Subjects randomized to receive active drug in study 165-302 part 2
- Pooled Placebo: Subjects randomized to receive placebo in study 165-302 part 2
Period: Overall Study
Arm/Group | Pooled Active | Pooled Placebo
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pooled Results: This is a sub-study of 165-302, with a randomized, placebo-control discontinuation design in Part 2. 9 subjects were enrolled in 165-303: 3 in 20mg/day and 3 in 40mg/day Active arm, 2 in 20mg/day and 1 in 40mg/day Placebo arm. Data interpretability was extremely limited, hence planned analysis was using the pooled treatment groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Active | Pooled Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.10) | 39.7 (9.24) | 31.9 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Rapid Visual Processing (RVP) Mean Response Latency (CANTAB Task)
Description: The RVP task measures sustained attention. In this task, a series of random digits continuously appears in the middle of the screen. Subjects are asked to recognize a specific sequence of digits and are asked to press a button on the screen whenever this specific sequence of digits appears within this series of continuous digits.
  RVP mean latency is the mean response latency during assessment sequence blocks where the subject responded correctly (Latency units are milliseconds). Lower scores represent better performance.
  Observed range for Pooled Active: -103.1 to 65.5 (change from baseline) Observed range for Pooled Placebo: -10.4 to 39.0 (change from baseline)
Time Frame: Baseline to Part 2 Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Millisec
Arm/Group | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 6 | 3
Millisec | -24.23 (60.161) | 18.03 (25.532)

2. Primary Outcome: Change From Baseline in Spatial Working Memory (SWM) Between Errors 4-8 Boxes (CANTAB Task)
Description: The SWM task measures visuospatial working memory. During this task, a number of boxes appears on a screen. The objective of the task is to find a token under a box and to place this token in a designated area. There is only one token under one box during each round and the location of the token rotates in each round to a different box, other than a box within which the token was found in previous rounds. The subject is therefore asked to remember which boxes previously contained tokens so as to better the chances and speed of finding tokens under boxes which did not previously contain tokens.
  SWM between errors measures the total number of times the subject revisits a box in which a token has previously been found in the same problem (calculated for assessed problems only).
  Observed range for Pooled Active: -8 to 1 (change from baseline) Observed range for Pooled Placebo: -5 to 12 (change from baseline)
  Lower scores represent better performance.
Time Frame: Baseline to Part 2 Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of times
Arm/Group | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 6 | 3
Number of times | -4.2 (3.06) | 3.0 (8.54)

3. Primary Outcome: Change From Baseline in Stop Signal Task (SST) Stop Signal Reaction T (CANTAB Task)
Description: The SST task measures inhibitory control and cognitive flexibility. The SST is a 2-part task. During part 1, an arrow appears on the screen and subjects are asked to press an arrow button on the screen corresponding with the direction of the arrow displayed. During part 2 of the task, subjects follow the same instructions as in part 1; however, they are asked to withhold their response (do not press an arrow button) if they hear an auditory signal (beep) when the arrow is displayed.
  SST stop signal delay is the length of time between the go stimulus and the stop stimulus at which the subject is able to successfully inhibit their response on 50% of trials. Lower time represents better performance.
  Observed range for Pooled Active: -31.6 to 48.7 (change from baseline) Observed range for Pooled Placebo: 47.8 to 72.5 (change from baseline)
Time Frame: Baseline to Part 2 Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Millisec
Arm/Group | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 6 | 3
Millisec | 8.42 (34.498) | 58.93 (12.529)

4. Secondary Outcome: Change From Baseline in RVP A Prime - Signal Detection Measure of Sensitivity to the Target (CANTAB Task)
Description: The RVP task measures sustained attention. In this task, a series of random digits continuously appears in the middle of the screen. Subjects are asked to recognize a specific sequence of digits and are asked to press a button on the screen whenever this specific sequence of digits appears within this series of continuous digits.
  RVP A prime represents the signal detection measure of sensitivity to the target, regardless of response tendency. In essence, measure of how good the subject is at detecting target sequences.
  Observed range for Pooled Active: -0.004 to 0.030 (change from baseline) Observed range for Pooled Placebo: -0.057 to -0.001 (change from baseline)
  A higher score on the test represents a better performance.
Time Frame: Baseline to Part 2 Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 6 | 3
Proportion | 0.0117 (0.01461) | -0.0247 (0.02899)

5. Secondary Outcome: Change From the Baseline in SWM Strategy 6-8 Boxes - Number of Distinct Boxes Used by the Subject to Begin a New Search for a Token(CANTAB Task)
Description: The SWM task measures visuospatial working memory. During this task, a number of boxes appears on a screen. The objective of the task is to find a token under a box and to place this token in a designated area. There is only one token under one box during each round and the location of the token rotates in each round to a different box, other than a box within which the token was found in previous rounds. The subject is therefore asked to remember which boxes previously contained tokens so as to better the chances and speed of finding tokens under boxes which did not previously contain tokens.
  For assessed problems with six boxes or more, SWM strategy is the number of distinct boxes used by the subject to begin a new search for a token (within the same problem). A high score represents poor use of this strategy and a low score equates to effective use.
  Observed range for Pooled Active: -3 to 3 (change from baseline) Observed range for Pooled Placebo: -3 to 1(change from baseline)
Time Frame: Baseline to Part 2 Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Number of distinct boxes
Arm/Group | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 6 | 3
Number of distinct boxes | -0.2 (2.32) | -1.0 (2.0)

6. Secondary Outcome: Change From Baseline in SST Proportion of Successful Stops - Measures the Proportion of Completed Stop Trials That Were Successful Stops (CANTAB Task)
Description: The SST task measures inhibitory control and cognitive flexibility. The SST is a 2-part task. During part 1, an arrow appears on the screen and subjects are asked to press an arrow button on the screen corresponding with the direction of the arrow displayed. During part 2 of the task, subjects follow the same instructions as in part 1; however, they are asked to withhold their response (do not press an arrow button) if they hear an auditory signal (beep) when the arrow is displayed. SST stop signal delay is the length of time between the go stimulus and the stop stimulus at which the subject is able to successfully inhibit their response on 50% of trials.
  SST proportion of successful stops measures the proportion of completed stop trials that were successful stops. A higher score on the test represents a better performance.
  Observed range for Pooled Active: -0.1 to 0.05 (change from baseline) Observed range for Pooled Placebo: 0.0 to 0.0 (change from baseline)
Time Frame: Baseline to Part 2 Week 8
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Pooled Active | Pooled Placebo
Number analyzed (Participants) | 6 | 3
Proportion | -0.0333 (0.04916) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: AE's were not monitored during this study (Adverse events were monitored through the parent 165-302 study (NCT01889862)), so this section is not applicable.
Description: Adverse Events were not collected as part of this observational sub study, but were reported to the parent 165-302 study
Arm/Group | Pooled Active | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT02468570/SAP_000.pdf
  • Study Protocol (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT02468570/Prot_001.pdf